CLINICAL TRIAL: NCT02323464
Title: Prevalence of Sleep Apnea in Patients Undergoing Surgery for Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Karl A Franklin (Other)
Responsible Party: Sponsor-Investigator, Karl A Franklin, Assoc prof, Umeå University
Organization: Umeå University (Other)
Other Study IDs: Dnr 2012-375-31M
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Sleep Apnea Syndromes; Hypoxia
MeSH Terms: conditions — Colorectal Neoplasms; Sleep Apnea Syndromes; Hypoxia | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Before surgery: patients scheduled for surgery of colorectal cancer
  Interventions: Procedure: Surgery for colorectal cancer
- Control subjects: Controls from the population without colorectal cancer
  Interventions: Other: No Interventions

INTERVENTIONS:
Procedure: Surgery for colorectal cancer — Includes open and minimally invasive surgery for colon- and rectal cancer
  Groups: Before surgery
Other: No Interventions — This is a control group from the population. They are not scheduled for surgery
  Groups: Control subjects

SUMMARY:
212 patients with colorectal cancer will be investigated before surgery and 100 of them after surgery. 597 individuals from a previous population based study will serve as controls to the prevalence of sleep apnea in the general population.

Investigations will include polysomonographic sleep apnea recordings during one night, lung function measurements, blood gas samples and questionnaires.

Controls: Men and women from two population-based cohort studies

DETAILED DESCRIPTION:
Inclusion: 212 patients with colorectal cancer will be investigated before surgery and 100 of them will also be investigated in the same manner after surgery. Due to drop-outs we calculate a need of inviting at least 250 patients.

Controls: 597 individuals from a previous population based study will serve as controls to the prevalence of sleep apnea in the general population.

Exclusion: Dementia, CPAP treated sleep apnea investigations: Patients are investigated with lung function, blood-gas samples, questionnaires, overnight polysomnographic sleep apnea recordings including oro-nasal airflow, thoraco-abdominal respiration belts, chin-EMG, EOG, EEG, ECG (V5) and body position.

Controls: Men and women from two population-based cohort studies the "Sleep and health in women" and the "Men in Uppsala: A Study of Sleep, Apnea and Cardiometabolic Health" and older men and women from a local senior organization.

Outcomes: Prevalence of sleep apnea and hypoxia, sleep quality, and lung function, blood gas, STOP-BANG, Epworth sleepiness scale, Mallampati score, symptoms of sleep apnea, surgical complications, mortality, cancer severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery of colorectal cancer

Exclusion Criteria:

* Dementia, CPAP treatment for obstructive sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery of colorectal cancer Healthy volunteers from population based studies will be included as controls
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of sleep apnea | 1 week
  Apnea-hypopnea index

SECONDARY OUTCOMES:
Sleep quality | 1 week
  total sleep time, sleep efficiency, time in different sleep stages
hypoxia, hypercapnia | 1 week
  blood-gas measurements
lung function | 1 week
  FVC, FEV1
subjective sleepiness | 1 week
  Eworth sleepiness scale
Mortality | Until death
  From the swedish death register
Side effects of surgery | 30 days
  From local register
Severity of cancer | 30 days
  Morphologic analysis of cancer type
nocturnal hypoxia | 1 week
  Pulsoximetry during polysomnography
Mallampati score | 1 day
  Inspection of mouth
STOP-Bang | 1 week
  Risk factor stratification
Symptoms of sleep apnea | 1 month
  snoring, daytime sleepiness, witnessed sleep apneas
Sex differences | 1 month
  Effect of sex on outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kar A Franklin, Ass prof, Principal Investigator — Dept of Surgical and perioperative sciences, Umeå University
Locations (1):
- Dept of Surgery, Inst of Surgical and Perioperative sciences, Umeå, Umea, Sweden